CLINICAL TRIAL: NCT02613728
Title: Accelerated Enhanced RECOVERy Following Minimally Invasive Colorectal Cancer Surgery (RecoverMI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Society of Colon and Rectal Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-0583; NCI-2016-00742 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-11-23; First posted 2015-11-24 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Colorectal cancer surgery; Polyp(s); Accelerated Enhanced Recovery; RecoverMI; Fluid diary; Questionnaires; Surveys; RecoverMI device
MeSH Terms: conditions — Colorectal Neoplasms; Polyps | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Arm (Active Comparator): Standard enhanced care following minimally invasive colorectal cancer surgery
  Interventions: Behavioral: Standard Enhanced Care
- Intervention (RecoverMI) Arm (Experimental): Routine care with Accelerated Recovery Plan, Early Discharge, and Telemedicine following minimally invasive colorectal cancer surgery
  Interventions: Behavioral: Accelerated Recovery Plan; Behavioral: Early Discharge; Other: Telemedicine

INTERVENTIONS:
Behavioral: Accelerated Recovery Plan
  Arms: Intervention (RecoverMI) Arm
Behavioral: Early Discharge
  Arms: Intervention (RecoverMI) Arm
Other: Telemedicine
  Arms: Intervention (RecoverMI) Arm
Behavioral: Standard Enhanced Care
  Arms: Standard of Care Arm

SUMMARY:
The goal of this clinical research study is to learn if RecoverMI care can help to shorten the time that patients are in the hospital after surgery and if it can help them recover sooner.

RecoverMI includes the following parts:

* Preoperative Education
* Early oral intake
* Early mobilization
* Telemedicine

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. This is done because no one knows if one group is the same, better, or worse than the other group.

* If you are assigned to Group 1, you will receive standard enhanced care after your surgery.
* If you are assigned to Group 2, you will receive routine care after surgery, but you will also receive accelerated recovery, early discharge, and Telemedicine. Participants will be loaned an iPad to use for video-conferencing and text messaging in this study.

This is an investigational study. The study doctor can explain how RecoverMI is designed to work.

Up to 32 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has histologically proven colorectal cancer or polyp(s) that is planned to be treated by surgical resection performed with curative intent.
2. Patient is >/= 18 years and younger than 80 years.
3. Elective minimally invasive operation.
4. No planned ostomy creation at time of enrollment.
5. Serum creatinine <1.5 measured within 30 days of surgery.
6. Ability to speak, read, and understand English.

Exclusion Criteria:

1. Strong, self-reported history of postoperative nausea and vomiting.
2. History of congestive heart failure. Systolic heart failure defined as Ejection Fraction (EF) </= 40%), or diastolic heart failure defined as EF >40% PLUS systemic manifestation of heart failure.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Cumulative Hospital Length of Stay (LOS) | 30 days post transplant

SECONDARY OUTCOMES:
Failure Rate (FR) in the RecoverMI Arm | 30 days
Patient Satisfaction | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: George Chang, MD, MS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Bednarski BK, Nickerson TP, You YN, Messick CA, Speer B, Gottumukkala V, Manandhar M, Weldon M, Dean EM, Qiao W, Wang X, Chang GJ. Randomized clinical trial of accelerated enhanced recovery after minimally invasive colorectal cancer surgery (RecoverMI trial). Br J Surg. 2019 Sep;106(10):1311-1318. doi: 10.1002/bjs.11223. Epub 2019 Jun 19. PMID 31216065
- [Derived] Price BA, Bednarski BK, You YN, Manandhar M, Dean EM, Alawadi ZM, Bryce Speer B, Gottumukkala V, Weldon M, Massey RL, Wang X, Qiao W, Chang GJ. Accelerated enhanced Recovery following Minimally Invasive colorectal cancer surgery (RecoverMI): a study protocol for a novel randomised controlled trial. BMJ Open. 2017 Jul 20;7(7):e015960. doi: 10.1136/bmjopen-2017-015960. PMID 28729319
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org